CLINICAL TRIAL: NCT02375113
Title: Soy as an Innovative Dietary Component in Abdominal Obesity Management
Brief Title: Soy as an Innovative Dietary Component in Abdominal Obesity Management Amongst Peri- and Early Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at San Antonio (Other)
Responsible Party: Principal Investigator, Dr. Meizi He, Professor, The University of Texas at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CRSGP 2012
Record Dates: First submitted 2013-02-28; First posted 2015-03-02 (Estimated); Results first posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2022-05

CONDITIONS: Central Obesity
Keywords: Obesity prevention; Soy supplementation
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Soy supplementation: Isoflavones 160 mg/day + 25 gram soy protein / day
  Interventions: Dietary Supplement: soy supplementation
- Control (Placebo Comparator): Placebo capsules + 25 gram whey protein / day
  Interventions: Dietary Supplement: soy supplementation

INTERVENTIONS:
Dietary Supplement: soy supplementation — Isoflavones will be in the form of capsule (80 mg /capsule). Placebo capsule will be filled with cellulose. These capsules will be identical in size and color. Soy protein will be prepared in the form of powder, containing 25 g of soy protein per package. Placebo powder will contain 25 g whole milk protein. Both powders will be available in vanilla and chocolate flavors, and look and taste similar. They could be mixed with water, milk and other beverages. Subjects will be asked to consume 2 capsules and 1 powder packet daily, preferably at breakfast for 6 months.
  Subjects failing to show up at the monthly visit for refilling supplement will be contacted by research staff via email or phone.

SUMMARY:
This is a pilot study examining the effect of dietary supplements that contain soy products. The purpose of this study to find out if soy supplementation can help to reduce the storage of a certain kind of fat on the body, visceral fat. Visceral fat is fat found deep in the abdomen; it has the potential to increase the risk of certain health problems.

DETAILED DESCRIPTION:
Obesity is a leading risk factor for many chronic diseases in the USA. Abdominal fat, specifically visceral fat is metabolically active and can be detrimental to health. Abdominal obesity is especially high in postmenopausal women (prevalence rates 50- 70%) in whom estrogen deficiency may lead to accumulation of excess visceral fat. Although estrogen replacement therapy is effective in preventing visceral fat accumulation, its adverse effects warrant a search for a safer phytochemical that exerts estrogenic properties. Soy, containing isoflavones (estrogen-like compounds), is a promising dietary component in reducing abdominal obesity in menopausal women. The favorable effects of isoflavones were already demonstrated in animal studies.The effects of soy compounds as a dietary component in preventing and reducing abdominal obesity and its associated metabolic abnormalities will be examined among menopausal Women. We will use quantitative magnetic resonance spectroscopy/imaging (qMRS/I) to determine dose and effects of soy supplementation for preventing and treating abdominal adiposity. The results from this study will shed light on the application of soy as a novel dietary approach in preventing and managing abdominal obesity among peri- and early menopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 45 and 60
2. experiencing irregular menses along with one or more other symptoms of menopause including: vaginal dryness, difficulty sleeping, hot flashes, mood changes, increased abdominal/belly fat, or with cessation of menstrual cycle for no more than three years
3. having a BMI greater than 25
4. Waist circumference greater than 88 cm
5. having the ability to understand study procedures and to comply with them for the entire length of the study.

Exclusion Criteria:

1. Have ever been diagnosed with cancer
2. Have tumors in the reproductive system
3. Allergies to soy or milk protein
4. Have known metabolic disorders that may affect body weight and body composition (e.g., hypercortisolism and hypothyroidism, non-alcoholic fatty liver disease)
5. Are receiving hormone replacement therapy or estrogen-like remedy
6. Are taking medications (e.g., thyroid, cortisol/cortisone, ephedra, thermogenics, etc) within 30 days prior to the start of the study.
7. Are emotional or uncontrolled eaters as measured by a brief screening tool Three-Factor Eating Questionnaire (TFEQ), i.e., 3 "yes" to the three emotional eating questions or 2 "yes" to the 2 uncontrolled eating questions.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meizi He, PhD, Principal Investigator — University of Texas at San Antonio
Locations (1):
- Human Nutrition Lab, UTSA, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after 12 months of study completion.
Access Criteria: Data access requests will be reviewed by an Review Panel at the University of Texas at San Antonio. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Result] Umana CK, Wilmoth S, Pan M, Zhang JQ, Fogt DL, He M. Effects of Soy Supplementation on Abdominal Obesity and Metabolic Risks on Post-Menopausal Women: A Pilot Study. Austin Journal of Obesity & Metabolic Syndrome. (1): 1-6, 2017.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a six-month randomized double-blind, placebo-controlled trial. Subjects, early post-menopausal women, were recruited from the local community via flyers, bulletin board advertisements and word-of-mouth referrals. Subjects were randomly assigned to either the Intervention group or the Control group .
Groups:
- Intervention: Soy supplementation: Isoflavones 160 mg/day + 25 gram soy protein / day
  soy supplementation: Isoflavones will be in the form of capsule (80 mg /capsule). Placebo capsule will be filled with cellulose. These capsules will be identical in size and color. Soy protein will be prepared in the form of powder, containing 25 g of soy protein per package. Placebo powder will contain 25 g whole milk protein. Both powders will be available in vanilla and chocolate flavors, and look and taste similar. They could be mixed with water, milk and other beverages. Subjects will be asked to consume 2 capsules and 1 powder packet daily, preferably at breakfast for 6 months.
  Subjects failing to show up at the monthly visit for refilling supplement will be contacted by research staff via email or phone.
- Control: Placebo capsules + 25 gram whey protein / day
  soy supplementation: Isoflavones will be in the form of capsule (80 mg /capsule). Placebo capsule will be filled with cellulose. These capsules will be identical in size and color. Soy protein will be prepared in the form of powder, containing 25 g of soy protein per package. Placebo powder will contain 25 g whole milk protein. Both powders will be available in vanilla and chocolate flavors, and look and taste similar. They could be mixed with water, milk and other beverages. Subjects will be asked to consume 2 capsules and 1 powder packet daily, preferably at breakfast for 6 months.
  Subjects failing to show up at the monthly visit for refilling supplement will be contacted by research staff via email or phone.
Period: Overall Study
Arm/Group | Intervention | Control
Started (Twelve met the inclusion criteria and consented to take part in the study.) | 6 (Six subjects were randomly assigned into Intervention.) | 6 (Six subjects were randomly assigned into Control.)
Completed | 4 | 4
Not Completed | 2 | 2
Not completed — Undisclosed Reason(s). | 1 | 1
Not completed — Poor adherence (<70%). | 1 | 0
Not completed — Discomfort of ingesting daily protein sh | 0 | 1

BASELINE CHARACTERISTICS:
Population: 12 subjects were randomly assigned into either Intervention or Control. 1 subject in the Control discontinued for undisclosed reasons; another dropped out due to ingestion discomfort; 1 Intervention subject discontinued for undisclosed reason. At study endpoint, 5 subjects remained in the Intervention, with 1 being excluded due to poor adherence.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (4.4) | 53.7 (4) | 54.0 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Body Fat (kg)
Description: Total body fat and abdominal fat were measured by DEXA (Hologic QDR Discovery A, Bedford, MA)
Time Frame: Study endpoint (6 months post intervention)
Population: The GLM Univariate procedure was used to determine intervention effects. The models included outcome measures as the dependent variable, treatment condition as the fixed factor (1=control; 2=intervention), and corresponding baseline outcome measures and age were covariates.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 4
kg
  Total body fat (kg) | 40.96 (0.84) | 40.12 (0.97)
  Abdominal fat (kg) | 2.94 (0.57) | 4.26 (0.49)

2. Secondary Outcome: BMI (kg/m^2)
Description: Body Mass Index (BMI) was calculated using the equation of weight (kg) over height (m) squared (kg/m^2)
Time Frame: Study endpoint (6 months post intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 4
kg/m^2 | 33.45 (0.5) | 33.64 (0.5)

3. Secondary Outcome: Blood Pressure (mmHg)
Description: Subjects' resting systolic and diastolic blood pressure (SBP and DBP, mmHg) was measured with an electronic sphygmomanometer (Omron, USA).
Time Frame: Study endpoint (6 months post intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 4
mm Hg
  SBP (mm Hg) | 125.41 (6.11) | 129.99 (6.64)
  DBP (mm Hg) | 73.06 (3.42) | 74.61 (3.55)

4. Secondary Outcome: Lipid Profile and Fasting Glucose
Description: High-density lipoprotein (HDL) (mg/L) normal range > 40 mg/dL Low-density lipoprotein (LDL) (mg/L) normal range <100 mg/dL Triglyceride (TG) (mg/L) normal range <150 mg/dl Fasting glucose (mg/dl) normal range: <100 mg/dl C-Reactive Protein (mg/dl): <3 mg/dl in healthy individuals
Time Frame: Study endpoint (6 months post intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 4
mg/dl
  TC (mg/dl) | 171.38 (3.45) | 175.16 (3.33)
  HDL (mg/dl) | 53.69 (3.13) | 47.66 (3.04)
  LDL (mg/dl) | 98.98 (6.42) | 106.9 (6.06)
  TG (mg/dl) | 114.05 (3.09) | 104.98 (3.19)
  Glucose (mg/dl) | 85.98 (2.08) | 89.47 (2.19)

5. Secondary Outcome: Waist Circumference (cm)
Description: Waist Circumference was measured midway between the iliac crest and bottom of the rib cage (cm)
Time Frame: Study endpoint (6 months post intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cm
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 4
cm | 105.59 (0.3) | 107.24 (0.3)

6. Secondary Outcome: Insulin Resistance
Description: Insulin sensitivity index as measured by homeostasis model assessment-insulin resistance (HOMA-IR Index): Normal range 0.5-1.4
Time Frame: Study endpoint (6 months post intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: HOMA-IR Index
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 4
HOMA-IR Index | 1.62 (0.42) | 1.62 (0.51)

7. Secondary Outcome: Inflammatory Cytokines IL-6 (ng/ml)
Description: Inflammatory cytokines IL-6 (ng/ml): 75-80 ng/ml in healthy individuals
Time Frame: Study endpoint (6 months post intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 4
ng/ml | 0.1 (0.05) | 0.04 (0.06)

8. Secondary Outcome: C-Reactive Protein (mg/L)
Description: C-Reactive Protein (mg/L) <3 mg/L in healthy individuals
Time Frame: Study endpoint (6 months post intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 4
mg/L | 3.11 (0.04) | 3.08 (0.05)

ADVERSE EVENTS:
Time Frame: The data and adverse effect was monitored from the start of the 6-month period to the end.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=6) | Control (N=6)
Discomfort of ingesting daily protein shake (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The small sample size led to insufficient statistical power to detect small intervention effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No